CLINICAL TRIAL: NCT06432907
Title: Decoding of Neuronal Potentials Associated With Motor Performance and Motor Imagery Obtained Using Intracranial stereoEEG Electrodes
Brief Title: StereoEEG Motor Neuronal Potentials Decoding
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Research Center of Neurology, Russia (Other Government)
Collaborators: Institute of Higher Nervous Activity and Neurophysiology of RAS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Stereo-iBCI
Record Dates: First submitted 2024-05-06; First posted 2024-05-29 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Drug Resistant Epilepsy; Brain-Computer Interfaces
Keywords: Brain-Computer Interface; Motor Imagery; Motor Performance; Intracranial Electroencephalography
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- StereoEEG (Experimental): Each patient will participate in one experimental session lasting no more than 60 minutes, recording brain signals associated with hand movement, motor imagery, and brain-computer interface (BCI) control.
  Interventions: Other: motor tasks

INTERVENTIONS:
Other: motor tasks — During the study session, the patient will sit at a table in front of a computer monitor. The stereoEEG electrodes will be connected to the Neurovisor-BMM52 electroencephalograph (Medical Computer Systems, Russia) and to a computer with a software for recording and decoding brain signals (BCI classifier). One microsensor (Ascension TrekStar, Ascension Technology, USA) and two disposable cutaneous electrodes (connected to the Neurovisor-BMM52 system) will be put on each patient's hand for electromyogram recording.
  The session consists from 3 blocks (1-3). The participant is asked to:
  1. execute simple motor tasks (thumbs up, open hand or clench hand into fist - 30 times with each hand with 5-second brakes), according to the instruction on the computer screen;
  2. to imagine the same movements - 30 times with each hand with 5-second brakes;
  3. to imagine the same movements with the feedback (brain-computer interface control).
  The blocks are separated by 5-minute brakes.
  Other Names: motor execution, motor imagery, brain-computer interface control with motor imagery paradigm

SUMMARY:
The goals of this study are (1) to evaluate the rate of stereoEEG brain-computer interface (BCI) classification accuracy and (2) to collect the dataset of neuronal signals recorded from stereoEEG electrodes during motor performance, motor imagery or brain-computer interface control. The study enrolls hospitalised patients suffering from resistant epilepsy with already implanted intracranial stereoEEG electrodes for medical reasons (i.e. for preoperative localization of the epileptogenic foci). The number and location of electrodes are determined solely for the clinical purposes of stereoEEG monitoring and are not related to the protocol of the current study.

After obtaining informed consent to participate in the study, each patient will participate in one experimental session lasting no more than 60 minutes, recording brain signals associated with hand movement, motor imagery, and BCI control. All tasks and instructions presented during the study session are not pro-epileptogenic and cannot provoke an epileptic attack. The experiments will take place in the patient's room, without interruption of observation by the department's medical staff.

The data recorded in this study will be used to improve or develop new algorithms for decoding motor signals from deep brain structures for their potential use in invasive BCIs.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients who have had stereoEEG electrodes implanted for medical reasons;
* voluntary informed consent to participate in the study;
* age from 18 to 70 years.

Exclusion Criteria:

* patient refusal to participate in the study;
* cognitive impairment that prevents following the study instructions;
* severe visual impairment that does not allow viewing visual instructions on a computer screen;
* upper limb paresis or other motor disorders;
* pain in the hand of any etiology;
* any acute diseases, exacerbation of chronic diseases, acute life-threatening conditions;
* occurrence of an epileptic attack during the experiment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Rate of BCI classification recall | During the procedure
  The proportion (%) of cases with correct identification of the task among all presentations of the corresponding command.

CONTACTS AND LOCATIONS:
Locations (1):
- Research center of neurology, Department of neurorehabilitation and physiotherapy, Moscow, Russia